CLINICAL TRIAL: NCT00493402
Title: The Efficacy, Safety, and Patient Reported Outcomes of Different Regimens of Transarterial Chemoembolization in Patients With Hepatocellular Carcinoma
Brief Title: Different Regimens of Transarterial Chemoembolization for Hepatocellular Carcinoma
Acronym: TACEforHCC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Ministry of Health, China (Other Government); Guangdong Provincial People's Hospital (Other); The 458 Hospital of Chinese PLA (Other); Kaiping Central Hospital (Other)
Responsible Party: Principal Investigator, Shi Ming, Dr., Sun Yat-sen University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: hcc-001
Record Dates: First submitted 2007-06-27; First posted 2007-06-28 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: Antineoplastic Agents; administration & dosage; Carcinoma, Hepatocellular; Chemoembolization, Therapeutic; Humans; Liver Neoplasms; therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- combined chemotherapy with embolization (Experimental): chemotherapy with lipiodol mixed with EADM 50mg, lobaplatin 50mg, and MMC 6mg, with particle embolization.
  Interventions: Procedure: Transarterial chemoembolization (TACE)
- combined chemotherapy without embolization (Experimental): chemotherapy with lipiodol mixed with EADM 50mg, lobaplatin 50mg, and MMC 6mg, without particle embolization.
  Interventions: Procedure: Transarterial chemoembolization (TACE)
- single agent chemotherapy with embolization (Experimental): chemotherapy with lipiodol mixed with EADM 50mg, plus particle embolization.
  Interventions: Procedure: Transarterial chemoembolization (TACE)

INTERVENTIONS:
Procedure: Transarterial chemoembolization (TACE) — drugs and dosage: chemotherapy with lipiodol mixed with EADM 50mg, lobaplatin 50mg, and MMC 6mg, plus particle embolization.
  Arms: combined chemotherapy with embolization
Procedure: Transarterial chemoembolization (TACE) — drugs and dosage: chemotherapy with lipiodol mixed with EADM 50mg, lobaplatin 50mg, and MMC 6mg.
  Arms: combined chemotherapy without embolization
Procedure: Transarterial chemoembolization (TACE) — Drugs and dosage:chemotherapy with lipiodol mixed with EADM 50mg, plus particle embolization.
  Arms: single agent chemotherapy with embolization

SUMMARY:
The purpose of this study is to evaluate efficacy, safety, and patient reported outcomes (PRO) of different regimens of transarterial chemoembolization (TACE) in patients with hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
Transarterial chemoembolization (TACE) has been recommended as first line non-curative therapy for non-surgical patients with large/multifocal HCC who do not have vascular invasion or extrahepatic spread. There has not been any standardized protocol in the choice of chemotherapeutic agents, dosage, dilution, rate of injection, and time interval between treatments. Similarly, there is no agreement on the choice of embolizing agents, degree of embolization, and whether the chemotherapeutic agent should be given together, or before the embolizing agent.

Comparison(s): In patients with HCC who underwent TACE therapy, stratified by whether they have vascular invasion and tumor size, we compare efficacy, safety, and patient reported outcomes (PRO) of different regimens of TACE.

Regimen 1: lipiodol combined chemotherapy with embolization

Regimen 2: lipiodol combined chemotherapy without embolization

Regimen 3: lipiodol single agent chemotherapy with embolization

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with minimal height of 150cm and minimal weight of 50 KG
* Histological confirmed HCC
* with no previous treatment
* With unresectable tumor
* With solitary or multiple intrahepatic tumor, the diameter of the largest one must larger than 7cm.
* No significant baseline liver dysfunction. Cirrhotic status of Child-Pugh class A only
* No significant renal impairment (creatinine clearance < 30 mL/minute)
* The following laboratory parameters:

  * Platelet count ≥ 60,000/µL
  * Hemoglobin ≥ 8.5 g/dL
  * Total bilirubin ≤ 1.5 mg/dL
  * ASL and AST ≤ 5 x upper limit of normal
  * Serum albumin ≥ 35 g/L
  * Serum creatinine ≤ 1.5 x upper limit of normal
  * INR ≤ 1.5 or a Pt/PTT within normal limits
  * Absolute neutrophil count (ANC) > 1,500/mm3
* Ability to understand the protocol and to agree to and sign a written informed consent document

Exclusion Criteria:

* Avascular tumor
* Main portal vein obstruction without cavernous transformation
* Evidence of hepatic decompensation including esophageal or gastric variceal bleeding or hepatic encephalopathy
* Obstructive jaundice
* Severe underlying cardiac or renal diseases
* Known or suspected allergy to the investigational agent or any agent given in association with this trial
* Pregnant or breast-feeding patients.
* History of organ allograft
* Active clinically serious infections
* Any condition that is unstable or which could jeopardize the safety of the patient and his/her compliance in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2007-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Overall survival | 3 years

SECONDARY OUTCOMES:
Time to progression | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Qing Li, M.D., Principal Investigator — Cancer Center, Sun Yat-set University
Locations (1):
- Cancer Center Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Bruix J, Sherman M; Practice Guidelines Committee, American Association for the Study of Liver Diseases. Management of hepatocellular carcinoma. Hepatology. 2005 Nov;42(5):1208-36. doi: 10.1002/hep.20933. No abstract available. PMID 16250051
- [Background] BREEDIS C, YOUNG G. The blood supply of neoplasms in the liver. Am J Pathol. 1954 Sep-Oct;30(5):969-77. No abstract available. PMID 13197542
- [Background] Llovet JM, Bruix J. Systematic review of randomized trials for unresectable hepatocellular carcinoma: Chemoembolization improves survival. Hepatology. 2003 Feb;37(2):429-42. doi: 10.1053/jhep.2003.50047. PMID 12540794
- [Background] Ono Y, Yoshimasu T, Ashikaga R, Inoue M, Shindou H, Fuji K, Araki Y, Nishimura Y. Long-term results of lipiodol-transcatheter arterial embolization with cisplatin or doxorubicin for unresectable hepatocellular carcinoma. Am J Clin Oncol. 2000 Dec;23(6):564-8. doi: 10.1097/00000421-200012000-00006. PMID 11202797
- [Background] Lau WY, Yu SC, Lai EC, Leung TW. Transarterial chemoembolization for hepatocellular carcinoma. J Am Coll Surg. 2006 Jan;202(1):155-68. doi: 10.1016/j.jamcollsurg.2005.06.263. Epub 2005 Oct 19. No abstract available. PMID 16377509
- [Background] Lopez PM, Villanueva A, Llovet JM. Systematic review: evidence-based management of hepatocellular carcinoma--an updated analysis of randomized controlled trials. Aliment Pharmacol Ther. 2006 Jun 1;23(11):1535-47. doi: 10.1111/j.1365-2036.2006.02932.x. PMID 16696801
- [Background] Lai CL, Wu PC, Chan GC, Lok AS, Lin HJ. Doxorubicin versus no antitumor therapy in inoperable hepatocellular carcinoma. A prospective randomized trial. Cancer. 1988 Aug 1;62(3):479-83. doi: 10.1002/1097-0142(19880801)62:33.0.co;2-l. PMID 2839280
- [Background] Hong K, Georgiades CS, Geschwind JF. Technology insight: Image-guided therapies for hepatocellular carcinoma--intra-arterial and ablative techniques. Nat Clin Pract Oncol. 2006 Jun;3(6):315-24. doi: 10.1038/ncponc0512. PMID 16757969
- [Background] Trevisani F, De Notariis S, Rossi C, Bernardi M. Randomized control trials on chemoembolization for hepatocellular carcinoma: is there room for new studies? J Clin Gastroenterol. 2001 May-Jun;32(5):383-9. doi: 10.1097/00004836-200105000-00005. PMID 11319307
- [Background] Kajanti M, Pyrhonen S, Mantyla M, Rissanen P. Intra-arterial and intravenous use of 4' epidoxorubicin combined with 5-fluorouracil in primary hepatocellular carcinoma. A randomized comparison. Am J Clin Oncol. 1992 Feb;15(1):37-40. doi: 10.1097/00000421-199202000-00008. PMID 1312770
- [Background] Heresbach D, Raoul JL, Bentue-Ferrer D, Bretagne JF, Van den Driessche J, Gastard J. [Chemotherapy combined with Lipiodol. In vitro study of the kinetics of release of adriamycin]. Gastroenterol Clin Biol. 1989 Oct;13(10):775-8. French. PMID 2556315
- [Background] Higashi S, Shimizu M, Nakashima T, Iwata K, Uchiyama F, Tateno S, Tamura S, Setoguchi T. Arterial-injection chemotherapy for hepatocellular carcinoma using monodispersed poppy-seed oil microdroplets containing fine aqueous vesicles of epirubicin. Initial medical application of a membrane-emulsification technique. Cancer. 1995 Mar 15;75(6):1245-54. doi: 10.1002/1097-0142(19950315)75:63.0.co;2-u. PMID 7882276
- [Background] Raoul JL, Heresbach D, Bretagne JF, Ferrer DB, Duvauferrier R, Bourguet P, Messner M, Gosselin M. Chemoembolization of hepatocellular carcinomas. A study of the biodistribution and pharmacokinetics of doxorubicin. Cancer. 1992 Aug 1;70(3):585-90. doi: 10.1002/1097-0142(19920801)70:33.0.co;2-#. PMID 1320447
- [Background] Kasugai H, Kojima J, Tatsuta M, Okuda S, Sasaki Y, Imaoka S, Fujita M, Ishiguro S. Treatment of hepatocellular carcinoma by transcatheter arterial embolization combined with intraarterial infusion of a mixture of cisplatin and ethiodized oil. Gastroenterology. 1989 Oct;97(4):965-71. doi: 10.1016/0016-5085(89)91505-9. PMID 2550311
- [Background] Nakao N, Uchida H, Kamino K, Nishimura Y, Ohishi H, Takayasu Y, Miura K. Determination of the optimum dose level of lipiodol in transcatheter arterial embolization of primary hepatocellular carcinoma based on retrospective multivariate analysis. Cardiovasc Intervent Radiol. 1994 Mar-Apr;17(2):76-80. doi: 10.1007/BF00193921. PMID 8013027
- [Background] Nakao N, Uchida H, Kamino K, Nishimura Y, Ohishi H, Takayasu Y, Nakamura H, Kuroda C, Fujita M, Yoshioka H, et al. Effectiveness of Lipiodol in transcatheter arterial embolization of hepatocellular carcinoma. Cancer Chemother Pharmacol. 1992;31 Suppl:S72-6. doi: 10.1007/BF00687110. PMID 1333913
- [Background] Takayasu K, Shima Y, Muramatsu Y, Moriyama N, Yamada T, Makuuchi M, Hasegawa H, Hirohashi S. Hepatocellular carcinoma: treatment with intraarterial iodized oil with and without chemotherapeutic agents. Radiology. 1987 May;163(2):345-51. doi: 10.1148/radiology.163.2.3031724.
- [Background] Nakamura H, Hashimoto T, Oi H, Sawada S. Transcatheter oily chemoembolization of hepatocellular carcinoma. Radiology. 1989 Mar;170(3 Pt 1):783-6. doi: 10.1148/radiology.170.3.2536946.
- [Background] Konno T. Targeting cancer chemotherapeutic agents by use of lipiodol contrast medium. Cancer. 1990 Nov 1;66(9):1897-903. doi: 10.1002/1097-0142(19901101)66:93.0.co;2-j. PMID 2171752
- [Background] Egawa H, Maki A, Mori K, Yamamoto Y, Mitsuhashi S, Bannai K, Asano K, Ozawa K. Effects of intra-arterial chemotherapy with a new lipophilic anticancer agent, estradiol-chlorambucil (KM2210), dissolved in lipiodol on experimental liver tumor in rats. J Surg Oncol. 1990 Jun;44(2):109-14. doi: 10.1002/jso.2930440210. PMID 2162452
- [Background] Mathupala SP, Rempel A, Pedersen PL. Glucose catabolism in cancer cells: identification and characterization of a marked activation response of the type II hexokinase gene to hypoxic conditions. J Biol Chem. 2001 Nov 16;276(46):43407-12. doi: 10.1074/jbc.M108181200. Epub 2001 Sep 13. PMID 11557773
- [Background] Ramsey DE, Kernagis LY, Soulen MC, Geschwind JF. Chemoembolization of hepatocellular carcinoma. J Vasc Interv Radiol. 2002 Sep;13(9 Pt 2):S211-21. doi: 10.1016/s1051-0443(07)61789-8. PMID 12354839
- [Background] Camma C, Schepis F, Orlando A, Albanese M, Shahied L, Trevisani F, Andreone P, Craxi A, Cottone M. Transarterial chemoembolization for unresectable hepatocellular carcinoma: meta-analysis of randomized controlled trials. Radiology. 2002 Jul;224(1):47-54. doi: 10.1148/radiol.2241011262. PMID 12091661
- [Background] Llovet JM, Real MI, Montana X, Planas R, Coll S, Aponte J, Ayuso C, Sala M, Muchart J, Sola R, Rodes J, Bruix J; Barcelona Liver Cancer Group. Arterial embolisation or chemoembolisation versus symptomatic treatment in patients with unresectable hepatocellular carcinoma: a randomised controlled trial. Lancet. 2002 May 18;359(9319):1734-9. doi: 10.1016/S0140-6736(02)08649-X. PMID 12049862
- [Background] Lo CM, Ngan H, Tso WK, Liu CL, Lam CM, Poon RT, Fan ST, Wong J. Randomized controlled trial of transarterial lipiodol chemoembolization for unresectable hepatocellular carcinoma. Hepatology. 2002 May;35(5):1164-71. doi: 10.1053/jhep.2002.33156. PMID 11981766
- [Background] Homma H, Mezawa S, Doi T, Miyanishi K, Takada K, Kukitsu T, Oku T, Masuko E, Nojiri S, Niitsu Y. A comparative randomized trial of intermittent intrahepatic arterial carboplatin- versus doxorubicin-lipiodol emulsion in advanced hepatocellular carcinoma (stage IV). Hepatogastroenterology. 2004 Jul-Aug;51(58):1135-9. PMID 15239261
- [Background] Stuart K. Chemoembolization in the management of liver tumors. Oncologist. 2003;8(5):425-37. doi: 10.1634/theoncologist.8-5-425. PMID 14530495
- [Background] Geschwind JF, Ramsey DE, Cleffken B, van der Wal BC, Kobeiter H, Juluru K, Hartnell GG, Choti MA. Transcatheter arterial chemoembolization of liver tumors: effects of embolization protocol on injectable volume of chemotherapy and subsequent arterial patency. Cardiovasc Intervent Radiol. 2003 Mar-Apr;26(2):111-7. doi: 10.1007/s00270-002-2524-6. Epub 2003 Mar 6. PMID 12616414